CLINICAL TRIAL: NCT06118853
Title: Impact of Yoga and Gentle Massage Practices on Symptom Management in Patients Undergoing Hematopoietic Stem Cell Transplantation at the Hospital Israelita Albert Einstein
Brief Title: Impact of Yoga and Gentle Massage Practices on Symptom Management in Patients Undergoing HSCT
Acronym: Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 61711022.6.0000.0071
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-11

CONDITIONS: Hematopoietic Stem Cell Transplantation; Bone Marrow Transplantation
Keywords: Hematopoietic Stem Cell Transplantation; Bone Marrow Transplantation; Integrative Therapies; Yoga; Massage
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups: Group A (control): standard treatment /Group B (intervention): yoga + gentle massage + standard treatment. Group B (intervention) will receive 8 individual integrative practice sessions at the bedside, each lasting 15 to 20 minutes, with 2 sessions per week during the following periods: from admission until D+0 / until D+7 / until D+14 / until D+21 or discharge. The therapist will choose the integrative practices that best suit the patient for each session, based on their psychophysical state and symptoms, as there can be many variations during HSCT. Group A (control) will receive 8 visits from integrative therapists who will remain in the patient's room, able to interact but without offering integrative practices, during the same periods described above. After D+21, these patients will also receive 8 integrative practice sessions at the bedside or in the Integrative Medicine room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control) (No Intervention): Standard treatment for HSCT
- Group B (intervention) (Experimental): Yoga or gentle massage plus standard treatment for HSCT
  Interventions: Behavioral: yoga or gentle massage plus standard treatment for HSCT

INTERVENTIONS:
Behavioral: yoga or gentle massage plus standard treatment for HSCT — The yoga sessions will be conducted at the patient's bedside, using one or more of the following techniques: gentle stretches (asanas), guided relaxation (savasana), slow and deep diaphragmatic breathing (pranayama), and meditative exercises focusing on natural breathing or visualization of a soothing place (dhyana). From these techniques, the integrative therapist will choose what best suits the patient for each session, based on their psychophysical state and symptoms presented, as there can be many variations during HSCT. Gentle massage is characterized by soft touches using light pressure, primarily using the palm of the hand, with a slow and steady rhythm across the entire body. It can be performed over clothing or even over the bedsheet and blanket.
  Arms: Group B (intervention)

SUMMARY:
This project aims to observe the impact of yoga and gentle massage practices on symptom management in patients undergoing Hematopoietic Stem Cell Transplantation (HSCT) at the Israelite Albert Einstein Hospital. It is a prospective, open label, randomized clinical study, comparing the practice of yoga or gentle massage combined with standard treatment versus standard treatment alone. Using the Edmonton Symptom Assessment System in 8 sessions, the investigators will analyze the domains of fatigue, pain, nausea, anxiety, and well-being before and after each session. The investigators will also assess Quality of Life - BMT, changes in Religiosity Scale before and after the intervention, and, at the end, Patient Satisfaction and subjective experience through a qualitative questionnaire. The hypothesis is that the practice of yoga and gentle massage combined with standard treatment is superior to standard treatment alone in symptom management in patients undergoing HSCT.

DETAILED DESCRIPTION:
Primary Objective: To assess the impact of yoga and/or gentle massage practices plus standard treatment versus standard treatment alone on symptom management in patients undergoing Hematopoietic Stem Cell Transplantation (HSCT), evaluated using the Edmonton Symptom Assessment Scale (ESAS).

Secondary Objectives:

* To analyze changes in the Quality-of-Life Scale during HSCT.
* To analyze changes in the Religiosity Scale during HSCT.
* To analyze the subjective experience of the patient during HSCT.
* To analyze patient satisfaction during HSCT. Hypothesis: The practice of yoga or gentle massage combined with standard treatment is superior to standard treatment alone in symptom management in patients undergoing HSCT.

Population: The study will be conducted at the Hospital Israelita Albert Einstein (HIAE), with patients admitted to the Oncology and Hematology Center for Bone Marrow Transplantation. Only after obtaining Informed Consent (IC) from the patient, clinical and sociodemographic variables during hospitalization will be extracted from the institutional electronic medical record database: age, gender, month/year and type of transplant, conditioning intensity, donor type, cell source, and underlying disease.

Inclusion Criteria: Adults aged 18 and above; admitted to HIAE, eligible for Bone Marrow Transplantation; patients who speak and read Portuguese.

Exclusion Criteria: Patients with hearing impairment; patients previously diagnosed with psychiatric disorders: schizophrenia.

Sample Size: The sample will consist of a minimum of 40 patients for this study.

Based on a pilot sample (n = 40) with only one session of yoga or gentle massage, a variation of 1.58 points (SD = 1.58 points) in fatigue improvement was observed. To find a mean difference of at least 1.5 points between the intervention group (yoga or gentle massage plus standard treatment) and the control group (standard treatment alone) in the proposed 8 sessions, with a power of 80% and a confidence level of 95%, the required sample size for the study would be 18 patients in each group. Since, in addition to fatigue, other parameters such as pain, nausea, anxiety, and well-being will also be evaluated, the investigators will use a sample of at least 20 patients per group to account for these parameters as well, totaling at least 40 patients in the study.

Randomization: Randomization will be carried out according to the randomization block generated by the Redcap tool. Therefore, upon agreeing to participate in the protocol, each patient will be entered into Redcap and randomized according to the specified parameters, stratified by age groups: 18 to 40 / 41 to 60 / above 61 years, and by type of transplant: autologous, allogeneic, and umbilical cord.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above;
* Admitted to HIAE, eligible for Bone Marrow Transplantation;
* Patients who speak and read the Portuguese language.

Exclusion Criteria:

* Patients with hearing impairment;
* Patients previously diagnosed with psychiatric disorder: schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Symptom Management: fatigue, pain, nausea, anxiety, and well-being | The sessions will occur at the following time points: Session 1 and 2 - from admission to Day 0 (infusion) / Session 3 and 4: between Day 1 and Day 7 / Session 5 and 6: between Day 8 and Day 14 / Session 7 and 8: between Day 15 and Day 21 or discharge.
  The Edmonton Symptom Assessment Scale will be administered both before and after each of the 8 sessions in both groups to evaluate pain, fatigue, nausea, anxiety, and well-being. The scale for each domain ranges from 0 to 10, where 0 signifies no symptoms or excellent well-being, and 10 signifies the most severe symptoms or worst possible well-being.

SECONDARY OUTCOMES:
Scale of Quality-of-Life | Two assessment points: upon admission and on Day 21 or at discharge (whichever comes first).
  The investigators will use the Functional Assessment Cancer Therapy - Bone Marrow Transplantation scale, which is a quality-of-life questionnaire designed to measure aspects of quality of life related to bone marrow transplantation. The scale ranges from 0, representing the worst possible quality of life or well-being, to 148, indicating the highest quality of life or well-being. This scale has been translated into Portuguese and validated for use in Brazilian patients.
Scale of Religiosity | Two assessment points: upon admission and on Day 21 or at discharge (whichever comes first).
  The Duke University Religion Index is a brief instrument for assessing aspects related to religiosity. The scale consists of five items that capture three dimensions of religiosity most related to health outcomes: organizational, non-organizational, and intrinsic religiosity. The score ranges from 1 to 27, with higher scores indicating greater religiosity. The scale has been translated into Portuguese and validated for use in Brazilian patients.
Qualitative Report | Day 21 or at discharge (whichever comes first).
  On Day 21, a Qualitative Report will be presented through RedCap, and patients will be invited to provide a written response to an open question: "How was your experience with Integrative Medicine?"
Patient-Reported Experience Measures | Day 21 or at discharge (whichever comes first).
  Investigators will utilize Patient-Reported Experience Measures with a scale ranging from 1 to 25, where higher scores indicate better patient experience and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Hamerschlak, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Maria Ester Azevedo Massola, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bazinet A, Popradi G. A general practitioner's guide to hematopoietic stem-cell transplantation. Curr Oncol. 2019 Jun;26(3):187-191. doi: 10.3747/co.26.5033. Epub 2019 Jun 1. PMID 31285665
- [Result] Gratwohl A, Baldomero H, Aljurf M, Pasquini MC, Bouzas LF, Yoshimi A, Szer J, Lipton J, Schwendener A, Gratwohl M, Frauendorfer K, Niederwieser D, Horowitz M, Kodera Y; Worldwide Network of Blood and Marrow Transplantation. Hematopoietic stem cell transplantation: a global perspective. JAMA. 2010 Apr 28;303(16):1617-24. doi: 10.1001/jama.2010.491. PMID 20424252
- [Result] Foord AM, Cushing-Haugen KL, Boeckh MJ, Carpenter PA, Flowers MED, Lee SJ, Leisenring WM, Mueller BA, Hill JA, Chow EJ. Late infectious complications in hematopoietic cell transplantation survivors: a population-based study. Blood Adv. 2020 Apr 14;4(7):1232-1241. doi: 10.1182/bloodadvances.2020001470. PMID 32227211
- [Result] Cohen MZ, Rozmus CL, Mendoza TR, Padhye NS, Neumann J, Gning I, Aleman A, Giralt S, Cleeland CS. Symptoms and quality of life in diverse patients undergoing hematopoietic stem cell transplantation. J Pain Symptom Manage. 2012 Aug;44(2):168-80. doi: 10.1016/j.jpainsymman.2011.08.011. Epub 2012 Jun 13. PMID 22699091
- [Result] Deng G. Integrative Medicine Therapies for Pain Management in Cancer Patients. Cancer J. 2019 Sep/Oct;25(5):343-348. doi: 10.1097/PPO.0000000000000399. PMID 31567462
- [Result] El-Jawahri A, LeBlanc T, VanDusen H, Traeger L, Greer JA, Pirl WF, Jackson VA, Telles J, Rhodes A, Spitzer TR, McAfee S, Chen YA, Lee SS, Temel JS. Effect of Inpatient Palliative Care on Quality of Life 2 Weeks After Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2016 Nov 22;316(20):2094-2103. doi: 10.1001/jama.2016.16786. PMID 27893130
- [Result] Grulke N, Albani C, Bailer H. Quality of life in patients before and after haematopoietic stem cell transplantation measured with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire QLQ-C30. Bone Marrow Transplant. 2012 Apr;47(4):473-82. doi: 10.1038/bmt.2011.107. Epub 2011 May 23. PMID 21602898
- [Result] Zetzl T, Renner A, Pittig A, Jentschke E, Roch C, van Oorschot B. Yoga effectively reduces fatigue and symptoms of depression in patients with different types of cancer. Support Care Cancer. 2021 Jun;29(6):2973-2982. doi: 10.1007/s00520-020-05794-2. Epub 2020 Oct 7. PMID 33026490
- [Result] Jim HS, Sutton SK, Jacobsen PB, Martin PJ, Flowers ME, Lee SJ. Risk factors for depression and fatigue among survivors of hematopoietic cell transplantation. Cancer. 2016 Apr 15;122(8):1290-7. doi: 10.1002/cncr.29877. Epub 2016 Jan 27. PMID 26814442
- [Result] Liang J, Lee SJ, Storer BE, Shaw BE, Chow EJ, Flowers ME, Krakow EF, Bar M, Syrjala KL, Salit RB, Kurukulasuriya CE, Jim HSL. Rates and Risk Factors for Post-Traumatic Stress Disorder Symptomatology among Adult Hematopoietic Cell Transplant Recipients and Their Informal Caregivers. Biol Blood Marrow Transplant. 2019 Jan;25(1):145-150. doi: 10.1016/j.bbmt.2018.08.002. Epub 2018 Aug 9. PMID 30098393
- [Result] Jeon M, Yoo IY, Kim S, Lee J. Post-traumatic growth in survivors of allogeneic hematopoietic stem cell transplantation. Psychooncology. 2015 Aug;24(8):871-7. doi: 10.1002/pon.3724. Epub 2014 Nov 10. PMID 25382562
- [Result] Corman M, Rubio MT, Cabrespine A, Brindel I, Bay JO, De La Tour RP, Dambrun M. Retrospective and prospective measures of post-traumatic growth reflect different processes: longitudinal evidence of greater decline than growth following a hematopoietic stem-cell transplantation. BMC Psychiatry. 2021 Jan 11;21(1):27. doi: 10.1186/s12888-020-03007-y. PMID 33430807
- [Result] Tick H, Nielsen A. Academic Consortium for Integrative Medicine & Health Commentary to Health and Human Services (HHS) on Inter-agency Task Force Pain Management Best Practices Draft Report. Glob Adv Health Med. 2019 Jul 17;8:2164956119857656. doi: 10.1177/2164956119857656. eCollection 2019. No abstract available. PMID 31360615
- [Result] Nakao M. Heart Rate Variability and Perceived Stress as Measurements of Relaxation Response. J Clin Med. 2019 Oct 16;8(10):1704. doi: 10.3390/jcm8101704. PMID 31623225
- [Result] Chen L, Michalsen A. Management of chronic pain using complementary and integrative medicine. BMJ. 2017 Apr 24;357:j1284. doi: 10.1136/bmj.j1284. PMID 28438745
- [Result] Hoffman JW, Benson H, Arns PA, Stainbrook GL, Landsberg GL, Young JB, Gill A. Reduced sympathetic nervous system responsivity associated with the relaxation response. Science. 1982 Jan 8;215(4529):190-2. doi: 10.1126/science.7031901.
- [Result] Mao JJ, Pillai GG, Andrade CJ, Ligibel JA, Basu P, Cohen L, Khan IA, Mustian KM, Puthiyedath R, Dhiman KS, Lao L, Ghelman R, Caceres Guido P, Lopez G, Gallego-Perez DF, Salicrup LA. Integrative oncology: Addressing the global challenges of cancer prevention and treatment. CA Cancer J Clin. 2022 Mar;72(2):144-164. doi: 10.3322/caac.21706. Epub 2021 Nov 9. PMID 34751943
- [Result] Witt CM, Balneaves LG, Cardoso MJ, Cohen L, Greenlee H, Johnstone P, Kucuk O, Mailman J, Mao JJ. A Comprehensive Definition for Integrative Oncology. J Natl Cancer Inst Monogr. 2017 Nov 1;2017(52). doi: 10.1093/jncimonographs/lgx012. PMID 29140493
- [Result] Lyman GH, Greenlee H, Bohlke K, Bao T, DeMichele AM, Deng GE, Fouladbakhsh JM, Gil B, Hershman DL, Mansfield S, Mussallem DM, Mustian KM, Price E, Rafte S, Cohen L. Integrative Therapies During and After Breast Cancer Treatment: ASCO Endorsement of the SIO Clinical Practice Guideline. J Clin Oncol. 2018 Sep 1;36(25):2647-2655. doi: 10.1200/JCO.2018.79.2721. Epub 2018 Jun 11. PMID 29889605
- [Result] Clarke TC, Barnes PM, Black LI, Stussman BJ, Nahin RL. Use of Yoga, Meditation, and Chiropractors Among U.S. Adults Aged 18 and Over. NCHS Data Brief. 2018 Nov;(325):1-8. PMID 30475686
- [Result] Cramer H, Lauche R, Langhorst J, Paul A, Michalsen A, Dobos G. Predictors of yoga use among internal medicine patients. BMC Complement Altern Med. 2013 Jul 13;13:172. doi: 10.1186/1472-6882-13-172. PMID 23849549
- [Result] Clarke TC, Black LI, Stussman BJ, Barnes PM, Nahin RL. Trends in the use of complementary health approaches among adults: United States, 2002-2012. Natl Health Stat Report. 2015 Feb 10;(79):1-16. PMID 25671660
- [Result] Kiecolt-Glaser JK, Bennett JM, Andridge R, Peng J, Shapiro CL, Malarkey WB, Emery CF, Layman R, Mrozek EE, Glaser R. Yoga's impact on inflammation, mood, and fatigue in breast cancer survivors: a randomized controlled trial. J Clin Oncol. 2014 Apr 1;32(10):1040-9. doi: 10.1200/JCO.2013.51.8860. Epub 2014 Jan 27. PMID 24470004
- [Result] Vadiraja HS, Raghavendra RM, Nagarathna R, Nagendra HR, Rekha M, Vanitha N, Gopinath KS, Srinath BS, Vishweshwara MS, Madhavi YS, Ajaikumar BS, Ramesh BS, Nalini R, Kumar V. Effects of a yoga program on cortisol rhythm and mood states in early breast cancer patients undergoing adjuvant radiotherapy: a randomized controlled trial. Integr Cancer Ther. 2009 Mar;8(1):37-46. doi: 10.1177/1534735409331456. Epub 2009 Feb 3. PMID 19190034
- [Result] Gonzalez M, Pascoe MC, Yang G, de Manincor M, Grant S, Lacey J, Firth J, Sarris J. Yoga for depression and anxiety symptoms in people with cancer: A systematic review and meta-analysis. Psychooncology. 2021 Aug;30(8):1196-1208. doi: 10.1002/pon.5671. Epub 2021 Mar 24. PMID 33763925
- [Result] McCall MC, Ward A, Heneghan C. Yoga in adult cancer: a pilot survey of attitudes and beliefs among oncologists. Curr Oncol. 2015 Feb;22(1):13-9. doi: 10.3747/co.22.2129. PMID 25684984
- [Result] Cramer H, Lauche R, Klose P, Lange S, Langhorst J, Dobos GJ. Yoga for improving health-related quality of life, mental health and cancer-related symptoms in women diagnosed with breast cancer. Cochrane Database Syst Rev. 2017 Jan 3;1(1):CD010802. doi: 10.1002/14651858.CD010802.pub2. PMID 28045199
- [Result] Swarm RA, Paice JA, Anghelescu DL, Are M, Bruce JY, Buga S, Chwistek M, Cleeland C, Craig D, Gafford E, Greenlee H, Hansen E, Kamal AH, Kamdar MM, LeGrand S, Mackey S, McDowell MR, Moryl N, Nabell LM, Nesbit S; BCPS; O'Connor N, Rabow MW, Rickerson E, Shatsky R, Sindt J, Urba SG, Youngwerth JM, Hammond LJ, Gurski LA. Adult Cancer Pain, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Aug 1;17(8):977-1007. doi: 10.6004/jnccn.2019.0038. PMID 31390582
- [Result] Cassileth BR, Vickers AJ. Massage therapy for symptom control: outcome study at a major cancer center. J Pain Symptom Manage. 2004 Sep;28(3):244-9. doi: 10.1016/j.jpainsymman.2003.12.016. PMID 15336336
- [Result] Mao JJ, Wagner KE, Seluzicki CM, Hugo A, Galindez LK, Sheaffer H, Fox KR. Integrating Oncology Massage Into Chemoinfusion Suites: A Program Evaluation. J Oncol Pract. 2017 Mar;13(3):e207-e216. doi: 10.1200/JOP.2016.015081. Epub 2017 Jan 3. PMID 28045616
- [Result] Shin ES, Seo KH, Lee SH, Jang JE, Jung YM, Kim MJ, Yeon JY. Massage with or without aromatherapy for symptom relief in people with cancer. Cochrane Database Syst Rev. 2016 Jun 3;2016(6):CD009873. doi: 10.1002/14651858.CD009873.pub3. PMID 27258432
- [Result] Boyd C, Crawford C, Paat CF, Price A, Xenakis L, Zhang W; Evidence for Massage Therapy (EMT) Working Group. The Impact of Massage Therapy on Function in Pain Populations-A Systematic Review and Meta-Analysis of Randomized Controlled Trials: Part II, Cancer Pain Populations. Pain Med. 2016 Aug;17(8):1553-1568. doi: 10.1093/pm/pnw100. Epub 2016 May 10. PMID 27165967
- [Result] Brandow AM, Carroll CP, Creary S, Edwards-Elliott R, Glassberg J, Hurley RW, Kutlar A, Seisa M, Stinson J, Strouse JJ, Yusuf F, Zempsky W, Lang E. American Society of Hematology 2020 guidelines for sickle cell disease: management of acute and chronic pain. Blood Adv. 2020 Jun 23;4(12):2656-2701. doi: 10.1182/bloodadvances.2020001851. PMID 32559294
- [Result] Bakshi N, Cooley A, Ross D, Hawkins L, Sullivan M, Astles R, Sinha C, Katoch D, Peddineni M, Gee BE, Lane PA, Krishnamurti L. A pilot study of the acceptability, feasibility and safety of yoga for chronic pain in sickle cell disease. Complement Ther Med. 2021 Jun;59:102722. doi: 10.1016/j.ctim.2021.102722. Epub 2021 Apr 21. PMID 33892094
- [Result] Ahles TA, Tope DM, Pinkson B, Walch S, Hann D, Whedon M, Dain B, Weiss JE, Mills L, Silberfarb PM. Massage therapy for patients undergoing autologous bone marrow transplantation. J Pain Symptom Manage. 1999 Sep;18(3):157-63. doi: 10.1016/s0885-3924(99)00061-5. PMID 10517036

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT06118853/Prot_000.pdf
  • Informed Consent Form (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT06118853/ICF_001.pdf